CLINICAL TRIAL: NCT03029637
Title: No-preparation Resin Bonded Bridges for the Replacement of Single Missing Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Michael G. Botelho, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 15-205a
Record Dates: First submitted 2016-12-30; First posted 2017-01-24 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Missing Teeth
Keywords: Resin bonded bridges; Randomized controlled trial
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No preparation resin bonded bridges (Experimental): RBBs with no or minimal preparation of their abutment teeth
  Interventions: Device: RBBs with no or minimal preparation of their abutment teeth
- Routine resin bonded bridges (Active Comparator): RBBs with routine tooth preparation of their abutment teeth
  Interventions: Device: RBBs with routine tooth preparation of their abutment teeth

INTERVENTIONS:
Device: RBBs with no or minimal preparation of their abutment teeth — Placement of resin bonded bridges on teeth with no or minimal cutting of their supporting teeth
  Arms: No preparation resin bonded bridges
Device: RBBs with routine tooth preparation of their abutment teeth — Placement of resin bonded bridges on teeth after routine cutting of their supporting teeth
  Arms: Routine resin bonded bridges

SUMMARY:
Tooth replacement is a significant issue in the World. Such replacement is considered important by patients to improve aesthetics, function and quality of life. Tooth replacement is therefore a significant issue. Resin-bonded bridges (RBBs) are conservative and cost-effective tooth replacement option that involves minimal tooth preparation and are secured in place with an adhesive cement by bonding to the outer enamel layer of the tooth. Clinical reports of these prostheses at the University of Hong Kong shows some of the highest success rate and greatest longevity in the dental literature. However, a problem with this type of prosthesis in that it still needs some tooth preparation to accommodate the framework thickness of the bridge. In some patients with tooth wear, this may mean cutting through the enamel crown down into dentine which will weaken the tooth. In light of the tooth preparation some patients will refuse this treatment, in particular patients with dental drill phobias.

The aim of this study is to investigate RBBs with tooth preparation and with no tooth preparation for the replacement of single missing teeth in a randomized controlled trial. However, a significant consequence of a no preparation RBB will mean that after cementation the prosthesis will interfere with the patient's bite, making the bridge prosthesis stand high. This will take time for the patient's original occlusion to re-establish itself by the movement of the tooth supporting the bridge. Despite the success of "supra-occluding" restoration has been reported in some studies, currently neither no preparation nor supraoccluding dental bridges are the standard of care for general dental practitioners and have not been reported on as a clinical trial in the literature. Most symptoms reported for supraoccluding restorations were transient and are reversible. The findings of this research will have significant impact on the teaching and practice for clinical prosthodontics and patient care worldwide. Patients will have a dental prosthesis that requires no dental drilling, no local anaesthetic and will have a stronger tooth supporting the bridge that should have greater longevity. More patients, in particular phobic patients will therefore seek treatment for tooth replacement with this conservative treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. 15+ years old
2. A complete bite on the supporting abutment tooth
3. At least one missing upper incisor
4. Controlled dental disease - no active caries or periodontal diseases
5. A minimum of 12 occluding pairs of natural teeth
6. Patients will be available to be clinically reviewed up to 3 years

Exclusion Criteria:

1. Patients with uncontrolled active tooth decay or periodontal disease (i.e. 5+ mm probing depth and bleeding on probing).
2. Patients with teeth missing opposite to the planned RBB
3. Abutment tooth mobility of 2 or greater (Millers classification)
4. Patients with debilitating illnesses or complicating medical conditions
5. Heavily restored tooth abutment not suitable for an RBB
6. A supporting abutment with an open bite

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prosthesis (resin bonded bridge RBB) retention/survival | 12 months
  Presence of the prosthesis in patient's mouth (Yes/No) by clinical visual examination
Prosthesis (resin bonded bridge RBB) retention/survival | 24 months
  Presence of the prosthesis in patient's mouth (Yes/No) by clinical visual examination
Prosthesis (resin bonded bridge RBB) retention/survival | 36 months
  Presence of the prosthesis in patient's mouth (Yes/No) by clinical visual examination

SECONDARY OUTCOMES:
Adverse events that related to no preparation/supra-occluding treatment approach | Up to 36 months
  Presence of clinical signs and symptoms or not (Yes/No) including but not limited to impact on patient's speech as well as thermal sensitivity, increased tooth mobility, periodontal/pulpal health of the abutment teeth
Time taken to re-establish the occlusion | Up to 36 months
  Settling of occlusion is judged by shimstock/occlusal marking paper on teeth adjacent to the prosthesis
Patient centered outcomes to the Prosthesis (I) | 36 months
  Subject's satisfaction (in visual analogue scale) on the RBB
Patient centered outcomes to the Prosthesis (II) | 36 months
  Impact of RBB on subject's oral health related quality of life (Oral Health Impact Profile, OHIP, in Likert scale)
Patient centered outcomes to the no preparation/supra-occluding treatment approach (I) | Up to 12 months
  Subject's satisfaction (in visual analogue scale) related to the no preparation/supraoccluding treatment approach RBBs
Patient centered outcomes to the no preparation/supra-occluding treatment approach (II) | Up to 12 months
  Impact of the no preparation/supraoccluding treatment approach on subject's oral health related quality of life (Oral Health Impact Profile, OHIP, in Likert scale)
Biomedical mediators of the no preparation/supra-occluding abutment teeth (I) | Up to 36 months
  Prostaglandin E2 level (pg/ul) in the gingival crevicular fluid of abutment teeth
Biomedical mediators of the contralateral control teeth (I) | Up to 36 months
  Prostaglandin E2 level (pg/ul) in the gingival crevicular fluid of contralateral control teeth
Biomedical mediators of the no preparation/supra-occluding abutment teeth (II) | Up to 36 months
  Human Interleukin-1 Family 2 level (pg/ul) in the gingival crevicular fluid of abutment teeth
Biomedical mediators of the contralateral control teeth (II) | Up to 36 months
  Human Interleukin-1 Family 2 level (pg/ul) in the gingival crevicular fluid of contralateral control teeth

CONTACTS AND LOCATIONS:
Locations (1):
- Prosthodontics, Faculty of Dentistry, The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No